CLINICAL TRIAL: NCT01250535
Title: Human Cytochrome P450 4F Enzymes and Drug Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kim Brouwer, PharmD, PhD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10-0576; 1R01GM089994-01A1 (NIH)
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Volunteers; Drug Drug Interactions
Keywords: Drug drug interactions; Warfarin; Anticoagulants; Lovastatin; Statins; CYP4F2; Vitamin K
MeSH Terms: interventions — Warfarin; Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin plus lovastatin (Experimental): Warfarin plus lovastatin
  Interventions: Drug: Warfarin; Drug: Lovastatin
- Warfarin plus placebo (Placebo Comparator): Warfarin plus placebo
  Interventions: Drug: Warfarin; Drug: Placebo

INTERVENTIONS:
Drug: Warfarin — 10 mg, po, single dose on day 7
  Other Names: Coumadin
Drug: Placebo — po, once a day, days 1 through 14
  Arms: Warfarin plus placebo
Drug: Lovastatin — 40 mg, po, once a day, days 1 through 14
  Other Names: Mevacor
  Arms: Warfarin plus lovastatin

SUMMARY:
Drug-drug interactions play an important role in clinical adverse events due to the prevalence of multi-drug therapy. Co-administration of warfarin and a statin has expanded substantially in the US over the last decades. The purpose of this study is to develop a mechanistic understanding of the role of a drug-metabolizing enzyme, CYP4F2, in the interaction between warfarin and statins. This study will test the hypothesis that lovastatin potentiates the anticoagulant effect of warfarin by inducing vitamin K-metabolizing enzyme CYP4F2 in humans, thus increasing warfarin's anticoagulant effect.

ELIGIBILITY:
Inclusion Criteria:

* Normal baseline clinical laboratory results including coagulation panel (prothrombin time (PT), international normalized ratio (INR), activated partial thromboplastin time (APTT)), liver function tests (ALT, AST, alkaline phosphatase and total bilirubin), kidney function tests (serum creatinine and BUN), lipid panel (cholesterol, LDL-C, HDL-C, and triglycerides), and blood creatine kinase
* Minimum weight of 110 lbs and minimum hemoglobin level at 12.5 g/dL
* Ability to understand the informed consent form
* Willing to abstain from grapefruit products, alcohol, and physical contact sports

Exclusion Criteria:

* History of intolerance, allergy, or hypersensitivity to study drugs warfarin and lovastatin or any substances contained in the medication
* History of clotting disorders, stroke, hypertension, anemia, renal insufficiency, hepatic dysfunction, platelet dysfunction, gastrointestinal bleeding, or any recent bleeding episode or trauma within 6 months
* History of significant medical conditions that the study physician believes would increase risk (e.g., additional bleeding disorders)
* Genotype non-homozygous for CYP2C9*1 or genotype VKORC1-1639AA
* History of significant alcohol abuse and/or illicit drug use
* Tobacco use within the month preceding the study
* Woman who is pregnant or breastfeeding
* Women who are unable to maintain adequate birth control during the study
* Post-menopausal women on estrogen replacement
* Chronic statin or warfarin use
* Taking concomitant medications, both prescription and non-prescription (including herbal products, over-the-counter medications, and multivitamins), known to alter lovastatin, warfarin, or vitamin K blood levels (women stabilized on hormonal methods of birth control will be allowed to participate, and subjects stabilized on antidepressant medications will be allowed to participate)
* Recent use of antibacterial antibiotics
* Recent blood donation or participation in other clinical studies within past 8 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics | Measurement will be performed before (baseline) and 2, 4, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, and 168h after co-administration of warfarin and lovastatin/placebo and during screening.
  Measurement of Prothrombin time (PT) to assess the International Normalized Ratio (INR).

SECONDARY OUTCOMES:
Pharmacokinetics | Sampling will be performed before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60, 72, 96, 120, 144, and 168 h after co-administration of warfarin and lovastatin/placebo.
  Vitamin K1 and vitamin K1 metabolite measured by maximum plasma concentration and AUC.
Pharmacokinetics | Sampling will be performed before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60, 72, 96, 120, 144, and 168 h after co-administration of warfarin and lovastatin/placebo.
  Pharmacokinetics for (R)- and (S)- Warfarin, and lovastatin measured by maximum plasma concentration and AUC.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Z Wang, PhD, Study Director — University of Kansas; Kim LR Brouwer, PharmD PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Clinical and Translational Research Center (CTRC), Chapel Hill, North Carolina, United States